CLINICAL TRIAL: NCT01519791
Title: A Multi-center, Randomized, Double-blind, Placebo-controlled Study to Evaluate the Efficacy and Safety of Certolizumab Pegol in Combination With Methotrexate for Inducing and Sustaining Clinical Response in the Treatment of DMARD-Naïve Adults With Early Active Rheumatoid Arthritis
Brief Title: A Multi-center, Randomized, Double-blind, Placebo-controlled Study to Evaluate the Efficacy and Safety of Certolizumab Pegol in Combination With Methotrexate in the Treatment of Disease Modifying Antirheumatic Drugs (DMARD)-naïve Adults With Early Active Rheumatoid Arthritis
Acronym: C-early
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UCB Pharma SA (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RA0055 Period 1; 2011-001729-25 (EudraCT Number)
Expanded Access: NCT03559686 (Available)
Record Dates: First submitted 2012-01-19; First posted 2012-01-27 (Estimated); Results first posted 2015-09-22 (Estimated); Last update posted 2018-07-31 (Actual); Status verified 2018-03

CONDITIONS: Rheumatoid Arthritis
Keywords: Certolizumab Pegol - Cimzia; Methotrexate; Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Certolizumab Pegol; Methotrexate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Certolizumab Pegol + Methotrexate (Experimental)
  Interventions: Biological: Certolizumab Pegol; Biological: Methotrexate
- Placebo + Methotrexate (Placebo Comparator)
  Interventions: Other: Placebo; Biological: Methotrexate

INTERVENTIONS:
Biological: Certolizumab Pegol — Prefilled syringes containing an injectable volume of 1 ml of solution for injection CZP for single use at a dosage strength of 200 mg/ml.
  Injections will be given subcutaneously. CZP 400 mg at Baseline, Week 2 and Week 4, followed by a maintenance dose of 200 mg every 2 Weeks until Week 50.
  Other Names: Cimzia; CZP
  Arms: Certolizumab Pegol + Methotrexate
Other: Placebo — 2 syringes Placebo at Baseline, Week 2 and Week 4, followed by 1 syringe Placebo every 2 Weeks.
  Arms: Placebo + Methotrexate
Biological: Methotrexate — The MTX treatment is to be initiated at a dose of 10 mg per Week (oral tablets at the strength of 2.5 mg/tablet). The MTX dosage should be escalated by 5 mg every 2 Weeks such that the maximum dosage of 25 mg per Week is achieved by Week 6 to Week 8. Patients who could not tolerate ≥ 15 mg/week MTX by Week 8 were withdrawn while the maximum tolerated dose per patient (optimized dose) was maintained to Week 52.
  Other Names: MTX

SUMMARY:
This study is intended to evaluate the efficacy and safety of Certolizumab Pegol (CZP) in combination with Methotrexate (MTX) for inducing and sustaining clinical response in the treatment of Disease Modifying Antirheumatic Drug (DMARD)-naïve adults with early active Rheumatoid Arthritis.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have a time since diagnosis of adult-onset Rheumatoid Arthritis (RA) less than 1 year as defined by the 2010 ACR/EULAR classification criteria from Screening Visit
* Positive Rheumatoid Factor (RF) and/or positive anticyclic Citrullinated Peptide Antibody (anti-CCP)
* Active RA disease
* DMARD-naïve
* Subject is naïve to RA related biologics

Exclusion Criteria:

* A diagnosis of any other inflammatory Arthritis
* History of infected joint prosthesis, or other significant infection and other serious medical condition
* Known Tuberculosis (TB) disease or high risk of acquiring TB infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 880 (Actual)
Dates: Start 2012-01; Primary Completion 2014-07 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — +1 877 822 9493 (UCB)
Locations (178):
- United States (70):
  - 209, Birmingham, Alabama
  - 170, Huntsville, Alabama
  - 180, Mobile, Alabama
  - 247, Glendale, Arizona
  - 165, Paradise Valley, Arizona
  - 234, Paradise Valley, Arizona
  - 243, Phoenix, Arizona
  - 251, Tucson, Arizona
  - 160, Covina, California
  - 257, Hemet, California
  - 159, Los Angeles, California
  - 201, San Leandro, California
  - 202, Upland, California
  - 172, Whittier, California
  - 190, Fort Lauderdale, Florida
  - 196, Jupiter, Florida
  - 238, Lake Mary, Florida
  - 232, Miami, Florida
  - 213, Naples, Florida
  - 214, Ocala, Florida
  - 237, Orange Park, Florida
  - 255, Orlando, Florida
  - 163, Palm Harbor, Florida
  - 166, Plantation, Florida
  - 192, Sarasota, Florida
  - 200, Vero Beach, Florida
  - 226, Coeur d'Alene, Idaho
  - 244, Springfield, Illinois
  - 224, South Bend, Indiana
  - 215, Cedar Rapids, Iowa
  - 191, Wichita, Kansas
  - 210, Wichita, Kansas
  - 177, Hagerstown, Maryland
  - 199, Kalamazoo, Michigan
  - 198, Eagan, Minnesota
  - 203, Tupelo, Mississippi
  - 179, St Louis, Missouri
  - 181, Lincoln, Nebraska
  - 256, Reno, Nevada
  - 229, Lebanon, New Hampshire
  - 228, Clifton, New Jersey
  - 207, Albuquerque, New Mexico
  - 176, Brooklyn, New York
  - 242, Plainview, New York
  - 227, Rochester, New York
  - 236, Durham, North Carolina
  - 245, Middleburg Heights, Ohio
  - 241, Oklahoma City, Oklahoma
  - 186, Portland, Oregon
  - 195, Bethlehem, Pennsylvania
  - 167, Duncansville, Pennsylvania
  - 168, Wyomissing, Pennsylvania
  - 189, Charleston, South Carolina
  - 205, Columbia, South Carolina
  - 204, Hendersonville, Tennessee
  - 217, Allen, Texas
  - 185, Amarillo, Texas
  - 161, Austin, Texas
  - 178, Corpus Christi, Texas
  - 162, Dallas, Texas
  - 184, Houston, Texas
  - 206, Houston, Texas
  - 223, Houston, Texas
  - 158, Mesquite, Texas
  - 175, Nassau Bay, Texas
  - 249, Plano, Texas
  - 197, San Antonio, Texas
  - 233, Kennewick, Washington
  - 183, Clarksburg, West Virginia
  - 174, Glendale, Wisconsin
- Argentina (4):
  - 276, Buenos Aires
  - 284, Rosario
  - 279, San Juan
  - 291, San Miguel de Tucumán
- Australia (8):
  - 6, Coffs Harbour, New South Wales
  - 2, Herson, Queensland
  - 1, Maroochydore, Queensland
  - 8, Woodville South, South Australia
  - 5, Fitzroy, Victoria
  - 4, Geelong, Victoria
  - 3, Malvern, Victoria
  - 7, Perth, Western Australia
- 50, Vienna, Austria
- Belgium (4):
  - 51, Brussels
  - 126, Gilly
  - 36, Kortrijk
  - 65, Yvoir
- Canada (4):
  - 240, Kelowna, British Columbia
  - 235, Hamilton, Ontario
  - 188, Montreal, Quebec
  - 194, Trois-Rivières, Quebec
- Colombia (8):
  - 303, Barranquilla
  - 272, Bogotá
  - 293, Bogotá
  - 299, Bogotá
  - 297, Bucaramanga
  - 288, Chía
  - 271, Medellín
  - 298, Medellín
- Czechia (4):
  - 108, Brno
  - 124, Bruntál
  - 38, Hradec Králové
  - 37, Prague
- France (5):
  - 16, Le Kremlin-Bicêtre
  - 85, Le Mans
  - 88, Montpellier
  - 34, Orléans
  - 79, Strasbourg
- Germany (16):
  - 52, Bad Doberan
  - 17, Bayreuth
  - 113, Berlin
  - 120, Berlin
  - 89, Erfurt
  - 70, Frankfurt
  - 71, Hamburg
  - 81, Hildesheim
  - 127, Lingen
  - 61, München
  - 53, Planegg
  - 132, Ratingen
  - 49, Rendsburg
  - 69, Rheine
  - 114, Würzburg
  - 59, Zerbst
- Hungary (6):
  - 18, Budapest
  - 21, Budapest
  - 86, Eger
  - 131, Szolnok
  - 110, Szombathely
  - 19, Veszprém
- Ireland (3):
  - 33, Cork
  - 54, Dublin
  - 32, Limerick
- Italy (5):
  - 115, Ferrara
  - 122, Milan
  - 40, Reggio Emilia
  - 72, Roma
  - 41, Verona
- Mexico (6):
  - 281, Durango
  - 286, Guadalajara
  - 292, Mexico City
  - 302, Mérida
  - 280, Monterrey
  - 294, San Luis Potosí City
- 78, Monaco, Monaco
- 42, Leiden, Netherlands
- Poland (7):
  - 128, Bydgoszcz
  - 67, Elblag
  - 99, Krakow
  - 92, Poznan
  - 74, Torun
  - 100, Warsaw
  - 44, Wroclaw
- Romania (7):
  - 58, Brasov
  - 111, Bucharest
  - 22, Bucharest
  - 25, Bucharest
  - 26, Bucharest
  - 24, Iași
  - 57, Lasi
- Spain (3):
  - 93, A Coruña
  - 47, Madrid
  - 63, Santiago de Compostela
- Sweden (6):
  - 76, Gothenburg
  - 82, Huddinge
  - 106, Lund
  - 123, Malmo
  - 77, Stockholm
  - 75, Uppsala
- Switzerland (2):
  - 118, Fribourg
  - 68, Sankt Gallen
- United Kingdom (7):
  - 125, Cannock
  - 105, Dudley
  - 56, Leeds
  - 121, London
  - 27, London
  - 80, Sheffield
  - 119, York

REFERENCES:
- [Result] Emery P, Bingham CO 3rd, Burmester GR, Bykerk VP, Furst DE, Mariette X, van der Heijde D, van Vollenhoven R, Arendt C, Mountian I, Purcaru O, Tatla D, VanLunen B, Weinblatt ME. Certolizumab pegol in combination with dose-optimised methotrexate in DMARD-naive patients with early, active rheumatoid arthritis with poor prognostic factors: 1-year results from C-EARLY, a randomised, double-blind, placebo-controlled phase III study. Ann Rheum Dis. 2017 Jan;76(1):96-104. doi: 10.1136/annrheumdis-2015-209057. Epub 2016 May 10. PMID 27165179
- [Result] Weinblatt ME, Bingham CO 3rd, Burmester GR, Bykerk VP, Furst DE, Mariette X, van der Heijde D, van Vollenhoven R, VanLunen B, Ecoffet C, Cioffi C, Emery P. A Phase III Study Evaluating Continuation, Tapering, and Withdrawal of Certolizumab Pegol After One Year of Therapy in Patients With Early Rheumatoid Arthritis. Arthritis Rheumatol. 2017 Oct;69(10):1937-1948. doi: 10.1002/art.40196. Epub 2017 Sep 12. PMID 28666080
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study started to enroll subjects in January 2012.
Pre-assignment Details: A total of 880 subjects were randomized. Three subjects were randomized in error, were not dosed, and withdrawn shortly afterwards as screen failures. Two of them were included in the Randomized Set 1 (RS1) only and one of these three subjects was conservatively excluded from any output. Therefore, 879 subjects are in RS1.
Groups:
- Placebo + Methotrexate: Placebo + Methotrexate (MTX)
  2 syringes Placebo at Baseline, Week 2 and Week 4 + MTX, followed by 1 syringe Placebo every 2 Weeks + MTX.
  The MTX treatment is to be initiated at a dose of 10 mg per Week. The MTX dosage should be escalated by 5 mg every 2 Weeks such that the maximum dosage of 25 mg per Week is achieved by Week 6 to Week 8.
- Certolizumab Pegol + Methotrexate: Certolizumab Pegol + Methotrexate (MTX)
  Prefilled syringes containing an injectable volume of 1 ml of solution for injection CZP for single use at a dosage strength of 200 mg/ml.
  Injections will be given subcutaneously. CZP 400 mg + MTX at Baseline, Week 2 and Week 4, followed by a maintenance dose of CZP 200 mg + MTX every 2 Weeks until Week 50.
  The MTX treatment is to be initiated at a dose of 10 mg per Week. The MTX dosage should be escalated by 5 mg every 2 Weeks such that the maximum dosage of 25 mg per Week is achieved by Week 6 to Week 8.
Period: Overall Study
Arm/Group | Placebo + Methotrexate | Certolizumab Pegol + Methotrexate
Started | 219 | 660
Completed Week 52 | 143 | 500
Completed | 67 | 292
Not Completed | 152 | 368
Not completed — SAE,non-fatal + AE,non-serious non-fatal | 2 | 1
Not completed — Protocol Violation | 6 | 19
Not completed — Other Reason | 87 | 222
Not completed — subjects randomized in error | 2 | 0
Not completed — Lack of Efficacy | 16 | 20
Not completed — SAE, non-fatal | 6 | 22
Not completed — AE, serious fatal | 0 | 1
Not completed — SAE, fatal + SAE, non-fatal | 0 | 1
Not completed — AE, non-serious non-fatal | 12 | 31
Not completed — Withdrawal by Subject | 15 | 37
Not completed — Lost to Follow-up | 6 | 14

BASELINE CHARACTERISTICS:
Population: Baseline Charactersitics refer to the Randomized Set (RS).
Arm/Group | Placebo + Methotrexate | Certolizumab Pegol + Methotrexate | Total Title
Number analyzed (Participants) | 219 | 660 | 879
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 2 | 3
  Between 18 and 65 years | 182 | 560 | 742
  >=65 years | 36 | 98 | 134
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.3 (13.2) | 50.5 (13.6) | 50.7 (13.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 175 | 499 | 674
  Male | 44 | 161 | 205

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects in Sustained Remission at Week 52
Description: Sustained remission is defined as a Disease Activity Score [Erythrocyte Sedimentation Rate] (DAS28[ESR]) < 2.6 at both Weeks 40 and 52.
  DAS28[ESR] is calculated using the Tender Joint Count (TJC), Swollen Joint Count (SJC) Erythrocyte Sedimentation Rate (ESR in mm/hour), and the Patient's Global Assessment of Disease Activity - Visual Analog Scale (PtGADA-VAS in mm) using the following formula:
  0.56 x √(TJC) + 0.28 x √(SJC) + 0.70 x lognat (ESR) + 0.014 x PtGADA, where 28 joints are examined and a lower score indicates less disease activity.
Time Frame: Week 52
Population: Full Analysis Set Period 1 (FAS1) with Non-Responder Imputation (NRI). FAS1 consisted of all subjects with valid Baseline and valid post-Baseline efficacy measurement within Period 1 for DAS28(ESR). For NRI, a subject having missing data for the time point assessed was conservatively counted as a nonremitter or nonresponder.
Measure: Number; unit: percentage of subjects
Groups:
- Placebo + Methotrexate (Full Analysis Set): Placebo + Methotrexate (MTX)
  2 syringes Placebo at Baseline, Week 2 and Week 4 + MTX, followed by 1 syringe Placebo every 2 Weeks + MTX.
  The MTX treatment is to be initiated at a dose of 10 mg per Week. The MTX dosage should be escalated by 5 mg every 2 Weeks such that the maximum dosage of 25 mg per Week is achieved by Week 6 to Week 8.
- Certolizumab Pegol + Methotrexate (Full Analysis Set): Certolizumab Pegol + Methotrexate (MTX)
  Prefilled syringes containing an injectable volume of 1 ml of solution for injection CZP for single use at a dosage strength of 200 mg/ml.
  Injections will be given subcutaneously. CZP 400 mg + MTX at Baseline, Week 2 and Week 4, followed by a maintenance dose of CZP 200 mg + MTX every 2 Weeks until Week 50.
  The MTX treatment is to be initiated at a dose of 10 mg per Week. The MTX dosage should be escalated by 5 mg every 2 Weeks such that the maximum dosage of 25 mg per Week is achieved by Week 6 to Week 8.
Arm/Group | Placebo + Methotrexate (Full Analysis Set) | Certolizumab Pegol + Methotrexate (Full Analysis Set)
Number analyzed (Participants) | 213 | 655
percentage of subjects | 15.0 | 28.9
Statistical Analysis 1: Comparison: Placebo + Methotrexate (Full Analysis Set) vs Certolizumab Pegol + Methotrexate (Full Analysis Set); In order to control the overall study-wise Type I error rate at 5 %, hypothesis testing was performed in the following hierarchical order (each at a 2-sided 95 % alpha level): 1. Primary: sustained DAS28(ESR) remission at Week 52 2. Key secondary: sustained DAS28(ESR) LDA at Week 52 3. ACR50 response at Week 52 in relation to Baseline 4. Change from Baseline in HAQ-DI at Week 52 5. Change from Baseline in mTSS at Week 52; Test type: Superiority or Other; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 2.283, 95% CI 2-sided [1.503 to 3.468] — The Odds ratio measuring the treatment effect was estimated from a logistic regression model including terms for treatment, region and stratification factor. Nonresponder imputation (NRI) was used

2. Secondary Outcome: Percentage of Subjects in Sustained Low Disease Activity (LDA) at Week 52
Description: Sustained LDA is defined as a Disease Activity Score [Erythrocyte Sedimentation Rate] (DAS28[ESR]) ≤ 3.2 at both Weeks 40 and 52.
Time Frame: Week 52
Population: as for outcome 1
Measure: Number; unit: percentage of subjects
Arm/Group | Placebo + Methotrexate (Full Analysis Set) | Certolizumab Pegol + Methotrexate (Full Analysis Set)
Number analyzed (Participants) | 213 | 655
percentage of subjects | 28.6 | 43.8
Statistical Analysis 1: Comparison: Placebo + Methotrexate (Full Analysis Set) vs Certolizumab Pegol + Methotrexate (Full Analysis Set); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 1.957, 95% CI 2-sided [1.384 to 2.767] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Change From Baseline in Modified Total Sharp Score (mTSS) to Week 52
Description: Van der Heijde modified Total Sharp Score (mTSS) is a methodology to assess the degree of joint damage by quantifying the extent of bone erosions and joint space narrowing for 44 and 42 joints, respectively. The mTSS ranges from 0 to 448, with higher scores representing greater damage.
Time Frame: From Baseline (Week 0) to Week 52
Population: The Radiographic Set Period 1 (RAD1) consisted of those subjects in the FAS1 who had provided valid radiographs (ie, radiographs resulting in a nonmissing mTSS score) at Baseline and at Week 52 or the Withdrawal Visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Placebo + Methotrexate (Radiographic Set): Placebo + Methotrexate (MTX)
  2 syringes Placebo at Baseline, Week 2 and Week 4 + MTX, followed by 1 syringe Placebo every 2 Weeks + MTX.
  The MTX treatment is to be initiated at a dose of 10 mg per Week. The MTX dosage should be escalated by 5 mg every 2 Weeks such that the maximum dosage of 25 mg per Week is achieved by Week 6 to Week 8.
- Certolizumab Pegol + Methotrexate (Radiographic Set): Certolizumab Pegol + Methotrexate (MTX)
  Prefilled syringes containing an injectable volume of 1 ml of solution for injection CZP for single use at a dosage strength of 200 mg/ml.
  Injections will be given subcutaneously. CZP 400 mg + MTX at Baseline, Week 2 and Week 4, followed by a maintenance dose of CZP 200 mg + MTX every 2 Weeks until Week 50.
  The MTX treatment is to be initiated at a dose of 10 mg per Week. The MTX dosage should be escalated by 5 mg every 2 Weeks such that the maximum dosage of 25 mg per Week is achieved by Week 6 to Week 8.
Arm/Group | Placebo + Methotrexate (Radiographic Set) | Certolizumab Pegol + Methotrexate (Radiographic Set)
Number analyzed (Participants) | 163 | 528
units on a scale | 1.8 (4.3) | 0.2 (3.2)
Statistical Analysis 1: Comparison: Placebo + Methotrexate (Radiographic Set) vs Certolizumab Pegol + Methotrexate (Radiographic Set); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA on ranks; Hodges-Lehmann point estimate of shift = -0.978, 95% CI 2-sided [-1.005 to -0.500] — ANCOVA model on the ranks with the terms for treatment, region, and time since RA diagnosis at Baseline (≤4 months or >4 months) as factors and rank Baseline value as a covariate. Confidence Interval is an asymptotic Moses CI

4. Secondary Outcome: Percentage of Subjects With Radiographic Non-progression From Baseline to Week 52
Description: Radiographic non-progression is defined as change in mTSS ≤ 0.5.
Time Frame: From Baseline (Week 0) to Week 52
Population: as for outcome 3
Measure: Number; unit: percentage of subjects
Arm/Group | Placebo + Methotrexate (Radiographic Set) | Certolizumab Pegol + Methotrexate (Radiographic Set)
Number analyzed (Participants) | 163 | 528
percentage of subjects | 49.7 | 70.3

5. Secondary Outcome: Change From Baseline in the Joint Erosion Score to Week 52
Description: Erosions were assessed in 16 locations per hand and 6 joints per foot. Erosions for each hand location were scored from 0 to 5, with 0 indicating no erosion. Scores 1 to 5 may have included combinations of discrete erosion(s) and/or large erosions. Erosions for each foot joint were scored from 0 to 10, with 0 indicating no erosions.
  The maximum possible erosion score for all 32-hand joints was 160. The maximum possible erosion score for all 12 feet joints was 120. Thus, the maximum possible total erosion score for hands and feet was 280.
Time Frame: From Baseline (Week 0) to Week 52
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo + Methotrexate (Radiographic Set) | Certolizumab Pegol + Methotrexate (Radiographic Set)
Number analyzed (Participants) | 163 | 528
units on a scale | 1.1 (3.0) | 0.1 (2.1)

6. Secondary Outcome: Change From Baseline in the Joint Narrowing Score to Week 52
Description: Joint space narrowing (JSN) was assessed in 15 locations per hand and 6 locations per foot. Joint space narrowing for each location was scored from 0 to 4, with 0 indicating no narrowing. The maximum possible score for JSN in all 30 hand joints was 120. The maximum possible score for JSN in all 12 feet joints was 48. Thus, the maximum possible total JSN score for Hands and feet was 168.
Time Frame: From Baseline (Week 0) to Week 52
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo + Methotrexate (Radiographic Set) | Certolizumab Pegol + Methotrexate (Radiographic Set)
Number analyzed (Participants) | 163 | 528
units on a scale | 0.7 (2.3) | 0.1 (1.7)

7. Secondary Outcome: Percentage of Subjects Meeting the American College of Rheumatology 20 % Response Criteria (ACR20) at Week 52
Description: The assessments are based on a 20 % or greater improvement from Baseline in the number of tender joints, a 20 % or more improvement in the number of swollen joints, and a 20% or greater improvement in 3 of the 5 remaining core set measures: Patient's Global Assessment of Disease Activity (PtGADA), Physician's Global Assessment of Disease Activity (PhGADA), Patient's Assessment of Arthritis Pain (PtAAP), physical function as assessed by the Health Assessment Questionnaire - Disability Index (HAQ-DI) and C-Reactive Protein (CRP).
Time Frame: From Baseline (Week 0) to Week 52
Population: as for outcome 1
Measure: Number; unit: percentage of subjects
Arm/Group | Placebo + Methotrexate (Full Analysis Set) | Certolizumab Pegol + Methotrexate (Full Analysis Set)
Number analyzed (Participants) | 213 | 655
percentage of subjects | 61.5 | 69.0

8. Secondary Outcome: Percentage of Subjects Meeting the American College of Rheumatology 50 % Response Criteria (ACR50) at Week 52
Description: The assessments are based on a 50 % or greater improvement from Baseline in the number of tender joints, a 50 %, or more improvement in the number of swollen joints, and a 50 % or greater improvement in 3 of the 5 remaining core set measures: Patient's Global Assessment of Disease Activity (PtGADA), Physician's Global Assessment of Disease Activity (PhGADA), Patient's Assessment of Arthritis Pain (PtAAP), physical function as assessed by the Health Assessment Questionnaire - Disability Index (HAQ-DI) and C-Reactive Protein (CRP).
Time Frame: From Baseline (Week 0) to Week 52
Population: as for outcome 1
Measure: Number; unit: percentage of subjects
Arm/Group | Placebo + Methotrexate (Full Analysis Set) | Certolizumab Pegol + Methotrexate (Full Analysis Set)
Number analyzed (Participants) | 213 | 655
percentage of subjects | 52.6 | 61.8
Statistical Analysis 1: Comparison: Placebo + Methotrexate (Full Analysis Set) vs Certolizumab Pegol + Methotrexate (Full Analysis Set); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.023, Regression, Logistic; Odds Ratio (OR) = 1.446, 95% CI 2-sided [1.052 to 1.989] — The Odds ratio was estimated from a logistic regression model including terms for treatment, region and stratification factor. Nonresponder imputation (NRI) was used

9. Secondary Outcome: Percentage of Subjects Meeting the American College of Rheumatology 70 % Response Criteria (ACR70) at Week 52
Description: The assessments are based on a 70 % or greater improvement from Baseline in the number of tender joints, a 70 %, or more improvement in the number of swollen joints, and a 70 % or greater improvement in 3 of the 5 remaining core set measures: Patient's Global Assessment of Disease Activity (PtGADA), Physician's Global Assessment of Disease Activity (PhGADA), Patient's Assessment of Arthritis Pain (PtAAP), physical function as assessed by the Health Assessment Questionnaire - Disability Index (HAQ-DI) and C-Reactive Protein (CRP).
Time Frame: From Baseline (Week 0) to Week 52
Population: as for outcome 1
Measure: Number; unit: percentage of subjects
Arm/Group | Placebo + Methotrexate (Full Analysis Set) | Certolizumab Pegol + Methotrexate (Full Analysis Set)
Number analyzed (Participants) | 213 | 655
percentage of subjects | 39.9 | 51.3

10. Secondary Outcome: Percentage of Subjects Meeting the 2011 American College of Rheumatology/ European League Against Rheumatism (ACR/EULAR) Remission Criteria at Week 52
Description: The ACR/EULAR 2011 remission criteria is defined as:
  Tender Joint Count (TJC) ≤ 1, Swollen Joint Count (SJC) ≤ 1, C-reactive protein (CRP) ≤ 1 mg/dl and Patient's Global Assessment of Disease Activity (PtGADA) ≤ 1.
Time Frame: Week 52
Population: as for outcome 1
Measure: Number; unit: percentage of subjects
Arm/Group | Placebo + Methotrexate (Full Analysis Set) | Certolizumab Pegol + Methotrexate (Full Analysis Set)
Number analyzed (Participants) | 213 | 655
percentage of subjects | 20.7 | 32.4

11. Secondary Outcome: Percentage of Subjects With Clinical Disease Activity Index (CDAI) ≤ 2.8 at Week 52
Description: CDAI is calculated as the sum of tender joint count (TJC), swollen joint count (SJC), Patient's Global Assessment of Disease Activity - Visual Analog Scale (PtGADA-VAS in mm), and Physician's Global Assessment of Disease Activity - Visual Analog Scale (PhGADA-VAS in mm). 28 joints are examined where a lower score indicates less disease activity.
Time Frame: Week 52
Population: as for outcome 1
Measure: Number; unit: percentage of subjects
Arm/Group | Placebo + Methotrexate (Full Analysis Set) | Certolizumab Pegol + Methotrexate (Full Analysis Set)
Number analyzed (Participants) | 213 | 655
percentage of subjects | 26.3 | 38.9

12. Secondary Outcome: Percentage of Subjects With Simplified Disease Activity Index (SDAI) ≤ 3.3 at Week 52
Description: SDAI is calculated as the sum of tender joint count (TJC), swollen joint count (SJC), Patient's Global Assessment of Disease Activity - Visual Analog Scale (PtGADA-VAS in mm), Physician's Global Assessment of Disease Activity - Visual Analog Scale (PhGADA-VAS in mm) and C-Reactive Protein (CRP in mg/L). 28 joints are examined where a lower score indicates less disease activity.
Time Frame: Week 52
Population: as for outcome 1
Measure: Number; unit: percentage of subjects
Arm/Group | Placebo + Methotrexate (Full Analysis Set) | Certolizumab Pegol + Methotrexate (Full Analysis Set)
Number analyzed (Participants) | 213 | 655
percentage of subjects | 24.9 | 38.9

13. Secondary Outcome: Percentage of Subjects With Disease Activity Score 28 [Erythrocyte Sedimentation Rate] (DAS28 [ESR]) < 2.6 at Week 52
Description: DAS28[ESR] is calculated using the Tender Joint Count (TJC), Swollen Joint Count (SJC) Erythrocyte Sedimentation Rate (ESR in mm/hour), and the Patient's Global Assessment of Disease Activity - Visual Analog Scale (PtGADA-VAS in mm) using the following formula:
  0.56 x √(TJC) + 0.28 x √(SJC) + 0.70 x lognat (ESR) + 0.014 x PtGADA, where 28 joints are examined and a lower score indicates less disease activity.
Time Frame: Week 52
Population: as for outcome 1
Measure: Number; unit: percentage of subjects
Arm/Group | Placebo + Methotrexate (Full Analysis Set) | Certolizumab Pegol + Methotrexate (Full Analysis Set)
Number analyzed (Participants) | 213 | 655
percentage of subjects | 26.8 | 42.6

14. Secondary Outcome: Percentage of Subjects Meeting the 2011 American College of Rheumatology/ European League Against Rheumatism (ACR/EULAR) Remission Criteria Simplified for Clinical Practice at Week 52
Description: The 2011 ACR/EULAR remission criteria simplified for clinical practice is defined as:
  Tender Joint Count (TJC) ≤ 1, Swollen Joint Count (SJC) ≤ 1 and Patient's Global Assessment of Disease Activity (PtGADA) ≤ 1.
Time Frame: Week 52
Population: as for outcome 1
Measure: Number; unit: percentage of subjects
Arm/Group | Placebo + Methotrexate (Full Analysis Set) | Certolizumab Pegol + Methotrexate (Full Analysis Set)
Number analyzed (Participants) | 213 | 655
percentage of subjects | 24.9 | 35.3

15. Secondary Outcome: Percentage of Subjects Achieving a Good or Moderate European League Against Rheumatism (EULAR) Response at Week 52
Description: Good response is defined as:
  DAS28[ESR] ≤ 3.2 and decrease from Baseline by > 1.2;
  moderate response is defined as achievement of one of the following:
  * DAS28[ESR] ≤ 3.2 and decrease from Baseline > 0.6 and ≤ 1.2
  * DAS28[ESR] > 3.2 and ≤ 5.1 and decrease from Baseline > 0.6
  * DAS28[ESR] > 5.1 and decrease from Baseline >1.2.
Time Frame: From Baseline (Week 0) to Week 52
Population: Full Analysis Set Period 1 (FAS1). The FAS1 consisted of all subjects who had a valid Baseline and valid post-Baseline efficacy measurement within Period 1 for the primary efficacy assessment of DAS28(ESR).
Measure: Number; unit: percentage of subjects
Arm/Group | Placebo + Methotrexate (Full Analysis Set) | Certolizumab Pegol + Methotrexate (Full Analysis Set)
Number analyzed (Participants) | 213 | 655
percentage of subjects | 82.2 | 89.9

16. Secondary Outcome: Change From Baseline in Disease Activity Score 28 [Erythrocyte Sedimentation Rate] (DAS28 [ESR]) to Week 52
Description: DAS28[ESR] is calculated using the Tender Joint Count (TJC), Swollen Joint Count (SJC) Erythrocyte Sedimentation Rate (ESR in mm/hour), and the Patient's Global Assessment of Disease Activity - Visual Analog Scale (PtGADA-VAS in mm) using the following formula:
  0.56 x √(TJC) + 0.28 x √(SJC) + 0.70 x lognat (ESR) + 0.014 x PtGADA, where 28 joints are examined and a lower score indicates less disease activity. A negative value in DAS28[ESR] change from Baseline indicates an improvement from Baseline.
Time Frame: From Baseline (Week 0) to Week 52
Population: Full Analysis Set Period 1 (FAS1) with Last Observation Carried Forward (LOCF). The FAS1 consisted of all subjects who had a valid Baseline and valid post-Baseline efficacy measurement within Period 1 for the primary efficacy assessment of DAS28(ESR). Missing DAS28(ESR) values were imputed using LOCF.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo + Methotrexate (Full Analysis Set) | Certolizumab Pegol + Methotrexate (Full Analysis Set)
Number analyzed (Participants) | 210 | 646
units on a scale | -3.014 (0.109) | -3.615 (0.069)

17. Secondary Outcome: Change From Baseline in Clinical Disease Activity Index (CDAI) to Week 52
Description: CDAI is calculated as the sum of tender joint count (TJC), swollen joint count (SJC), Patient's Global Assessment of Disease Activity - Visual Analog Scale (PtGADA-VAS in mm), and Physician's Global Assessment of Disease Activity - Visual Analog Scale (PhGADA-VAS in mm). 28 joints are examined where a lower score indicates less disease activity.
  The CDAI score ranges from 0 to 76, with a negative value in CDAI change from Baseline indicating an improvement from Baseline.
Time Frame: From Baseline (Week 0) to Week 52
Population: Full Analysis Set Period 1 (FAS1) with Last Observation Carried Forward (LOCF). The FAS1 consisted of all subjects who had a valid Baseline and valid post-Baseline efficacy measurement within Period 1 for the primary efficacy assessment of DAS28(ESR). Missing CDAI values were imputed using LOCF.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo + Methotrexate (Full Analysis Set) | Certolizumab Pegol + Methotrexate (Full Analysis Set)
Number analyzed (Participants) | 210 | 644
units on a scale | -29.09 (0.84) | -33.11 (0.52)

18. Secondary Outcome: Change From Baseline in Simplified Disease Activity Index (SDAI) to Week 52
Description: SDAI is calculated as the sum of tender joint count (TJC), swollen joint count (SJC), Patient's Global Assessment of Disease Activity - Visual Analog Scale (PtGADA-VAS in mm), Physician's Global Assessment of Disease Activity - Visual Analog Scale (PhGADA-VAS in mm) and C-Reactive Protein (CRP in mg/L). 28 joints are examined where a lower score indicates less disease activity.
  The SDAI score ranges from 0 to 86, with a negative value in SDAI change from Baseline indicating an improvement from Baseline.
Time Frame: From Baseline (Week 0) to Week 52
Population: Full Analysis Set Period 1 (FAS1) with Last Observation Carried Forward (LOCF). The FAS1 consisted of all subjects who had a valid Baseline and valid post-Baseline efficacy measurement within Period 1 for the primary efficacy assessment of DAS28(ESR). Missing SDAI values were imputed using LOCF.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo + Methotrexate (Full Analysis Set) | Certolizumab Pegol + Methotrexate (Full Analysis Set)
Number analyzed (Participants) | 210 | 644
units on a scale | -30.24 (0.88) | -34.55 (0.55)

19. Secondary Outcome: Percentage of Subjects With a Health Assessment Questionnaire- Disability Index (HAQ-DI) ≤ 0.5 at Week 52
Description: Normative physical function is defined as HAQ-DI score ≤ 0.5. The domains of the HAQ-DI are dressing and grooming, arising, eating, walking, hygiene, reach, grip and common daily activities.
  The total score ranges from 0 to 3 with lower scores meaning lower disability.
Time Frame: Week 52
Population: as for outcome 1
Measure: Number; unit: percentage of subjects
Arm/Group | Placebo + Methotrexate (Full Analysis Set) | Certolizumab Pegol + Methotrexate (Full Analysis Set)
Number analyzed (Participants) | 213 | 655
percentage of subjects | 35.7 | 48.1

20. Secondary Outcome: Change From Baseline in the Health Assessment Questionnaire - Disability Index (HAQ-DI) to Week 52
Description: The domains of the HAQ-DI are dressing and grooming, arising, eating, walking, hygiene, reach, grip and common daily activities.
  The total score ranges from 0 (no difficulty) to 3 (unable to do) with lower scores meaning lower disability.
  A negative value in HAQ-DI change from Baseline indicates an improvement from Baseline.
Time Frame: From Baseline (Week 0) to Week 52
Population: Full Analysis Set Period 1 (FAS1) with Last Observation Carried Forward (LOCF). The FAS1 consisted of all subjects who had a valid Baseline and valid post-Baseline efficacy measurement within Period 1 for the primary efficacy assessment of DAS28(ESR). Missing HAQ-DI values were imputed using LOCF.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo + Methotrexate (Full Analysis Set) | Certolizumab Pegol + Methotrexate (Full Analysis Set)
Number analyzed (Participants) | 210 | 645
units on a scale | -0.819 (0.044) | -0.997 (0.028)
Statistical Analysis 1: Comparison: Placebo + Methotrexate (Full Analysis Set) vs Certolizumab Pegol + Methotrexate (Full Analysis Set); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA; Difference in Least Squares (LS) Means = -0.177, 95% CI 2-sided [-0.273 to -0.082], Standard Error of Mean 0.049 — The CfB in HAQ-DI at Week 52 was analyzed using an ANCOVA model with terms for treatment, region, and time since Rheumatoid Arthritis (RA) diagnosis at Baseline (≤4 months or >4 months) as factors and Baseline value as a covariate

21. Secondary Outcome: Change From Baseline in the Bristol Rheumatoid Arthritis Fatigue- Multidimensional Questionnaire (BRAF-MDQ) Total Score to Week 52
Description: BRAF-MDQ total score ranges from 0 to 70 (with higher scores indicating worse fatigue).
  A negative value in BRAF-MDQ change from Baseline indicates an improvement from Baseline.
Time Frame: From Baseline (Week 0) to Week 52
Population: Full Analysis Set Period 1 (FAS1) with Last Observation Carried Forward (LOCF). The FAS1 consisted of all subjects who had a valid Baseline and valid post-Baseline efficacy measurement within Period 1 for the primary efficacy assessment of DAS28(ESR). Missing BRAF-MDQ values were imputed using LOCF.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo + Methotrexate (Full Analysis Set) | Certolizumab Pegol + Methotrexate (Full Analysis Set)
Number analyzed (Participants) | 205 | 636
units on a scale | -15.6 (1.0) | -17.8 (0.6)

22. Secondary Outcome: Number of Work Days Missed (Work Productivity Survey - Rheumatoid Arthritis [WPS-RA]) at Week 52
Description: Number of work days missed in the last month for employed subjects.
Time Frame: Week 52
Population: Full Analysis Set Period 1 (FAS1) with Last Observation Carried Forward (LOCF). The FAS1 consisted of all subjects who had a valid Baseline and valid post-Baseline efficacy measurement within Period 1 for the primary efficacy assessment of DAS28(ESR). Missing WPS-RA values were imputed using LOCF.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Placebo + Methotrexate (Full Analysis Set) | Certolizumab Pegol + Methotrexate (Full Analysis Set)
Number analyzed (Participants) | 106 | 351
days | 0.9 (2.5) | 0.6 (2.6)

23. Secondary Outcome: Number of Work Days With Reduced Productivity (Work Productivity Survey - Rheumatoid Arthritis [WPS-RA]) at Week 52
Description: Number of work days with reduced productivity in the last month for employed subjects.
Time Frame: Week 52
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Placebo + Methotrexate (Full Analysis Set) | Certolizumab Pegol + Methotrexate (Full Analysis Set)
Number analyzed (Participants) | 106 | 351
days | 1.8 (4.7) | 1.0 (3.4)

24. Secondary Outcome: Interference With Work Productivity (Work Productivity Survey - Rheumatoid Arthritis [WPS-RA]) at Week 52
Description: The Arthritis interference in the last month with work productivity is measured on a scale that ranges from 0 (no interference) to 10 (complete interference) for employed subjects.
Time Frame: Week 52
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo + Methotrexate (Full Analysis Set) | Certolizumab Pegol + Methotrexate (Full Analysis Set)
Number analyzed (Participants) | 106 | 351
units on a scale | 1.9 (2.3) | 1.4 (2.0)

25. Secondary Outcome: Number of Days With no Household Work (Work Productivity Survey - Rheumatoid Arthritis [WPS-RA]) at Week 52
Description: Number of days with no household work in the last month.
Time Frame: Week 52
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Placebo + Methotrexate (Full Analysis Set) | Certolizumab Pegol + Methotrexate (Full Analysis Set)
Number analyzed (Participants) | 206 | 640
days | 3.0 (6.7) | 1.9 (5.1)

26. Secondary Outcome: Number of Days With Reduced Household Work Productivity (Work Productivity Survey - Rheumatoid Arthritis [WPS-RA]) at Week 52
Description: Number of days with reduced household work productivity in the last month.
Time Frame: Week 52
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Placebo + Methotrexate (Full Analysis Set) | Certolizumab Pegol + Methotrexate (Full Analysis Set)
Number analyzed (Participants) | 206 | 640
days | 3.0 (6.6) | 2.1 (5.3)

27. Secondary Outcome: Number of Days With Hired Outside Help (Work Productivity Survey - Rheumatoid Arthritis [WPS-RA]) at Week 52
Description: Number of days with hired outside help in the last month.
Time Frame: Week 52
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Placebo + Methotrexate (Full Analysis Set) | Certolizumab Pegol + Methotrexate (Full Analysis Set)
Number analyzed (Participants) | 206 | 640
days | 0.7 (3.3) | 0.6 (3.2)

28. Secondary Outcome: Number of Days Missed of Family/Social/Leisure Activities (Work Productivity Survey - Rheumatoid Arthritis [WPS-RA]) at Week 52
Description: Number of days missed of family/social/leisure activities in the last month.
Time Frame: Week 52
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Placebo + Methotrexate (Full Analysis Set) | Certolizumab Pegol + Methotrexate (Full Analysis Set)
Number analyzed (Participants) | 206 | 640
days | 0.9 (3.1) | 0.9 (3.6)

29. Secondary Outcome: Interference With Household Work Productivity (Work Productivity Survey - Rheumatoid Arthritis [WPS-RA]) at Week 52
Description: The Arthritis interference in the last month with household work productivity is measured on a scale that ranges from 0 (no interference) to 10 (complete interference).
Time Frame: Week 52
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo + Methotrexate (Full Analysis Set) | Certolizumab Pegol + Methotrexate (Full Analysis Set)
Number analyzed (Participants) | 206 | 640
units on a scale | 2.5 (2.8) | 1.9 (2.5)

30. Secondary Outcome: Percentage of Subjects Achieving Low Disease Activity (LDA) at Week 52
Description: LDA is defined as achieving a Disease Activity Score 28 [Erythrocyte Sedimentation Rate] (DAS28 [ESR]) ≤ 3.2.
Time Frame: Week 52
Population: as for outcome 1
Measure: Number; unit: percentage of subjects
Arm/Group | Placebo + Methotrexate (Full Analysis Set) | Certolizumab Pegol + Methotrexate (Full Analysis Set)
Number analyzed (Participants) | 213 | 655
percentage of subjects | 39.4 | 54.7

ADVERSE EVENTS:
Time Frame: Adverse Events were collected from Screening over Baseline (Week 0) and Treatment Period 1 (Week 2 to Week 52) to the Safety Follow-Up Visit (Week 60).
Description: Adverse Events presented below refer to the Safety Set 1 (SS1), which consisted of all subjects in the Randomized Set who had received at least 1 dose of study medication (CZP/PBO) in Period 1.
Arm/Group | Placebo + Methotrexate | Certolizumab Pegol + Methotrexate
Serious Adverse Events (participants affected / at risk) | 20/217 | 70/659
Other Adverse Events (participants affected / at risk) | 63/217 | 248/659
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo + Methotrexate (N=217) | Certolizumab Pegol + Methotrexate (N=659)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 3 (5)
Bone marrow toxicity (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 1 (1)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac tamponade (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 1 (1)
Pericarditis (Cardiac disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Duodenal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Erosive duodenitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastritis erosive (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mesenteric panniculitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Bile duct stone (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 2 (2)
Anaphylactic shock (Immune system disorders) | 0 (0) | 1 (1)
Food allergy (Immune system disorders) | 0 (0) | 1 (1)
Abscess limb (Infections and infestations) | 0 (0) | 1 (1)
Appendiceal abscess (Infections and infestations) | 0 (0) | 1 (1)
Arthritis infective (Infections and infestations) | 0 (0) | 1 (1)
Breast abscess (Infections and infestations) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1)
Bronchopneumonia (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 2 (2)
Erysipelas (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Groin abscess (Infections and infestations) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1)
Impetigo (Infections and infestations) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 1 (1)
Kidney infection (Infections and infestations) | 0 (0) | 1 (1)
Labyrinthitis (Infections and infestations) | 1 (1) | 0 (0)
Latent tuberculosis (Infections and infestations) | 2 (2) | 1 (1)
Localised infection (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 3 (3) | 4 (4)
Pulmonary tuberculosis (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Staphylococcal infection (Infections and infestations) | 0 (0) | 1 (1)
Tuberculosis gastrointestinal (Infections and infestations) | 0 (0) | 1 (1)
Urosepsis (Infections and infestations) | 0 (0) | 1 (1)
Wound infection (Infections and infestations) | 0 (0) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (2)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Tendon rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Lupus-like syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (4)
Rheumatoid nodule (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Chondrosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Carpal tunnel syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 1 (1)
Cervicobrachial syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 1 (1)
Loss of consciousness (Nervous system disorders) | 0 (0) | 1 (1)
Migraine (Nervous system disorders) | 0 (0) | 1 (1)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Bladder outlet obstruction (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1) | 1 (1)
Menorrhagia (Reproductive system and breast disorders) | 0 (0) | 2 (4)
Uterine polyp (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Epiglottic cyst (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Laryngeal polyp (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (3)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Coronary arterial stent insertion (Surgical and medical procedures) | 0 (0) | 1 (1)
Hip arthroplasty (Surgical and medical procedures) | 0 (0) | 1 (1)
Leg amputation (Surgical and medical procedures) | 0 (0) | 1 (2)
Aortic aneurysm (Vascular disorders) | 0 (0) | 1 (1)
Aortic stenosis (Vascular disorders) | 0 (0) | 1 (1)
Arteriosclerosis (Vascular disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo + Methotrexate (N=217) | Certolizumab Pegol + Methotrexate (N=659)
Nausea (Gastrointestinal disorders) | 22 (22) | 83 (92)
Upper respiratory tract infection (Infections and infestations) | 11 (12) | 72 (86)
Urinary tract infection (Infections and infestations) | 16 (18) | 48 (63)
Nasopharyngitis (Infections and infestations) | 13 (17) | 46 (60)
Alanine aminotransferase increased (Investigations) | 9 (13) | 42 (46)
Headache (Nervous system disorders) | 8 (11) | 45 (65)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days